CLINICAL TRIAL: NCT06417346
Title: Comparison of Laparoscopic and Open Inguinal Hernia Repair in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Eşref Ulutaş (Other)
Collaborators: Van Training and Research Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Mehmet Eşref Ulutaş, Principal Investigator, Konya City Hospital
Organization: Konya City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65646564
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Urinary Retention; Postoperative Complications; Pain; Relapse
MeSH Terms: conditions — Urinary Retention; Postoperative Complications; Pain; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic TEP Repair under General Anesthesia (Experimental): A mini-incision was made at the umbilical margin, passing through the skin and subcutaneous tissue to expose the external sheath of the rectus muscle. The RS was incised, and the rectus muscle was laterally displaced. A 10-mm trocar was inserted into the preperitoneal space, and CO2 insufflation was performed with a pressure set at 12 mmHg. Two additional 5 mm trocars were inserted between the umbilicus and the symphysis pubis under laparoscopic guidance. Using laparoscopic dissectors and graspers, all steps of myopectineal orifice dissection were performed (16). A 15 × 10 cm prolene mesh was spread and secured to cover both direct and indirect hernia areas, extending approximately 2-3 cm beyond. Trocars were removed under camera surveillance after CO2 desufflation, and the skin was closed.
  Interventions: Procedure: Laparoscopic TEP Repair
- Open Technique (Lichtenstein) under Spinal Anesthesia (Active Comparator): Following a classic inguinal incision of approximately 5-7 cm extending laterally from the pubic tubercle, the external oblique aponeurosis was opened, the external ring was disrupted, and the spermatic cord/round ligament was suspended. The hernia sac was isolated from surrounding tissues and the spermatic cord/round ligament, then either reduced or ligated. Subsequently, a polypropylene mesh measuring approximately 60x110 mm² was placed to completely cover the transverse fascia, and continuous sutures were used to secure it laterally along the transverse arch starting from the pubic tubercle. Hemostasis was achieved, and the layers and skin were anatomically closed.
  Interventions: Procedure: Open Technique (Lichtenstein)

INTERVENTIONS:
Procedure: Laparoscopic TEP Repair — Laparoscopic TEP Repair performed
  Arms: Laparoscopic TEP Repair under General Anesthesia
Procedure: Open Technique (Lichtenstein) — Open Technique (Lichtenstein) performed
  Arms: Open Technique (Lichtenstein) under Spinal Anesthesia

SUMMARY:
Inguinal hernia is one of the most frequently performed surgeries in general surgery. This surgery can be performed with both open and laparoscopic techniques. There is no clear consensus on whether inguinal hernia repair, which is one of the most frequently performed surgeries in elderly patients, should be performed open or laparoscopic. The application of the open technique with regional anesthesia methods such as spinal anesthesia and local anesthesia makes these methods attractive. The fact that laparoscopic techniques cause patients to recover faster also makes these techniques attractive. However, the fact that it is usually performed under general anesthesia is a significant disadvantage. Increasing comorbidities and increased drug use, especially in elderly patients, make surgeons think about which technique to prefer. The aim of this study is to compare open and laparoscopic inguinal hernia repair, which should be preferred in patients over 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inguinal hernias.
* Patients aged over 65.

Exclusion Criteria:

* Younger than 65 years.
* Incarcerated or strangulated inguinal hernias.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-06-04 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
rate of postoperative mortality | postoperative 24 hours

SECONDARY OUTCOMES:
rate of urinary retansion | postoperative 24 hours
rate of postoperative pain | postoperative 24 hours
Rate of Hernia recurrence | first year
Rate of Postoperative complications | postoperative 24 hours and 1st month
  such as wound infection, bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science Van Training and Research Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vigneswaran Y, Gitelis M, Lapin B, Denham W, Linn J, Carbray J, Ujiki M. Elderly and octogenarian cohort: Comparable outcomes with nonelderly cohort after open or laparoscopic inguinal hernia repairs. Surgery. 2015 Oct;158(4):1137-43; discussion 1143-4. doi: 10.1016/j.surg.2015.08.002. Epub 2015 Aug 20. PMID 26299283
- [Result] Xi S, Chen Z, Lu Q, Liu C, Xu L, Lu C, Cheng R. Comparison of laparoscopic and open inguinal-hernia repair in elderly patients: the experience of two comprehensive medical centers over 10 years. Hernia. 2024 Aug;28(4):1195-1203. doi: 10.1007/s10029-024-03004-0. Epub 2024 Apr 4. PMID 38573484
- [Result] Bowling K, El-Badawy S, Massri E, Rait J, Atkinson J, Leong S, Stuart A, Srinivas G. Laparoscopic and open inguinal hernia repair: Patient reported outcomes in the elderly from a single centre - A prospective cohort study. Ann Med Surg (Lond). 2017 Aug 29;22:12-15. doi: 10.1016/j.amsu.2017.08.013. eCollection 2017 Oct. PMID 28878892
- [Derived] Ulutas ME, Yilmaz AH. Comparison of open and laparoscopic inguinal hernia repair in the elderly patients: a randomized controlled trial. Hernia. 2025 May 23;29(1):179. doi: 10.1007/s10029-025-03368-x. PMID 40407912